CLINICAL TRIAL: NCT03215446
Title: Evaluation of Total (Pre and Post) Conditioning on Rhabdomyolysis of Sedation With Sevoflurane Versus Propofol in Vascular Surgery With Clamping
Brief Title: Evaluate the Muscle Protection Effect of Sevoflurane Sedation in Vascular Surgery
Acronym: PHAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STEINBERG-GIRARD 2015
Record Dates: First submitted 2017-06-26; First posted 2017-07-12 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Vascular Surgery
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol (Active Comparator)
  Interventions: Drug: maintenance of anaesthesia with propofol
- sevoflurane (Experimental)
  Interventions: Drug: maintenance of anaesthesia with sevoflurane

INTERVENTIONS:
Drug: maintenance of anaesthesia with propofol
  Arms: propofol
Drug: maintenance of anaesthesia with sevoflurane
  Arms: sevoflurane

SUMMARY:
Halogenated anaesthetic agents (HAA) may induce protective processes by pre-conditioning the myocardium. All of the literature shows that HAA induce pre-conditioning, thanks to a class effect, and Sevoflurane is the most widely used today.

In humans, the protective effects of halogenated agents have principally been studied in heart surgery and have shown encouraging clinical results. It seems that HAA induce both pre-conditioning of the myocardium (early and late) and post conditioning.

Given these protective effects of HAA, in 2007, the American Heart Association (AHA) recommended the use of HAA for anaesthesia maintenance in non-cardiac surgery in patients with a high cardio-vascular risk. The aim of this study is to show a decrease in rhabdomyolysis and tissue distress (kidneys, myocardium and liver), thanks to Sevoflurane anaesthesia, in the post-operative period following vascular surgery with clamping

ELIGIBILITY:
Inclusion Criteria:

* persons who have provided written consent
* patients over 18 years of age
* patients undergoing scheduled vascular surgery with high clamping for:
* Abdominal aortic aneurysm
* suprapopliteal vascular bypass (aorto-bi-femoral, femoral trifurcation, ilio-femoral or femoro-femoral, femoro-popliteal).

Exclusion Criteria:

* persons without health insurance cover
* patients younger than 18 years of age, pregnant or breast-feeding women and adults under guardianship
* patients with epilepsy
* emergency surgery
* patient presenting a contra-indication for Sevoflurane: hypersensitivity to sevoflurane or to other halogenated anaesthetic agents, myopathy, hyper-eosinophilia, immunoallergic hepatitis, known or suspected genetic predisposition to malignant hyperthermia
* patients presenting a contra-indication to the use of Propofol: known hypersensitivity to propofol or to one of the constituents of the product, allergy to peanuts or soja
* Patients presenting a contra-indication for sufentanil: hypersensitivity to sufentanil or to opioids
* Association with opioid agonists-antagonists or partial opioid antagonists
* patients presenting a CI for the use of Cisatracurium: history of allergy or hypersensitivity to cisatracurium or atracurium
* patients presenting cardiac, respiratory, renal or kidney failure, hypovolemia, poor general health
* Patients with a risl of prolongation of the QT interval
* Patients with end-stage renal failure - requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
change from baseline Creatine PhosphoKinase | up to 24 hours post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No